CLINICAL TRIAL: NCT02347930
Title: Establish and Apply the Evaluation System of Ultrasonic Integrated Technology for Prevention and Treatment of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014DFT30090
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; ultrasound technology
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — only plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Confirmed acute kidney injury: Confirmed acute kidney injury
  Interventions: Other: kidney ultrasound

INTERVENTIONS:
Other: kidney ultrasound — kidney ultrasound

SUMMARY:
Establish an integrated evaluation system of ultrasound technology for the prognosis of acute kidney injury, and in order to achieve non-invasive, reliable early diagnosis "gold standard". Set up collabration with the expert in National Cheng Kung University Medical Center of Taiwan who did a lot of excellent work in basic research of prevention the progression of acut kidney injury. Study the experience about prevention progression of kidney disease in clinical and basic field. Establish cooperation with the professional in Hong Kong University of Science and Technology. To set up the system of natural products research and assess the Astragalus medicinal value.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. Clinical diagnosis of acute or chronic kidney injury
  2. Male or female, aged 18-80 years old
  3. signed informed consent
  4. Patients can breathe in, breathe out and hold their breathe with ease, communication without difficulty.

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Refuse to sign informed consent
  2. allergy to micro bubble hexafluoride drug
  3. Patients with cardiopulmonary insufficiency, pleural effusion, pulmonary infections
  4. Patients with asthma, chronic bronchitis
  5. Patients with pregnancy
  6. Patients can't cooperate or have a difficulty in breathing in, breathing out or holding their breathe
  7. Patients beening diagnosed with End-stage kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed acute kidney injury
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-04; Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
compare the results of kidney ultrasound with biomarkers of acute kidney injury | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: shan mou, Dr., Principal Investigator — Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of nephrology , Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China